CLINICAL TRIAL: NCT05467982
Title: Brief Intervention to Increase COVID-19 Knowledge in People With Serious Mental Illness
Brief Title: Brief COVID-19 Intervention for People With Serious Mental Illness and Co-Morbid Medical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sarah Pratt, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00031245
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Mental Illness; Chronic Disease
Keywords: integrated health; mental health; illness management; cardiovascular disease; physical health
MeSH Terms: conditions — Mental Disorders; Chronic Disease; Psychological Well-Being; Cardiovascular Diseases | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT: (Experimental): In addition to the primary intervention (Integrated Illness Management and Recovery), participants received 3 additional COVID-19 related educational/skills training sessions provided individually, remotely by I-IMR Specialists.
  Interventions: Behavioral: Integrated Illness Management and Recovery
- Stanford Chronic Disease Self-Management Program (CDSMP) ONLY: (Experimental): No additional COVID-19 intervention was provided to this group. These participants only received the primary disease management intervention (CDSMP)
  Interventions: Behavioral: Chronic Disease Self-Management Program

INTERVENTIONS:
Behavioral: Integrated Illness Management and Recovery — Education and skills training groups on illness management of chronic medical and psychiatric illness. Subsample of 75 will also receive COVID-specific Integrated Illness Management and Recovery module.
  Arms: Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT:
Behavioral: Chronic Disease Self-Management Program — Education and skills training groups on illness management of chronic conditions
  Arms: Stanford Chronic Disease Self-Management Program (CDSMP) ONLY:

SUMMARY:
The study will enroll 600 people with serious mental illness who receive services at Centerstone in KY or TN and will compare two different evidence-based self-management interventions: Integrated Illness Management and Recovery (I-IMR), a program developed by the study team at Dartmouth that trains people with serious mental illness on physical and mental health self-management, and the Stanford Chronic Disease Self-Management Program (CDSMP), a program largely focused on physical health self-management that has been used widely in the general population. In addition, PCORI is funding an evaluation of a COVID-related intervention that will begin in the Fall 2020.

DETAILED DESCRIPTION:
The proposed study will be the first to compare two commonly used but substantially different, evidence-based self-management interventions. Integrated Illness Management and Recovery (I-IMR), is an individually-tailored, 16-session, integrated program combining both physical and mental health self-management specifically developed for people with SMI. In contrast, the Stanford Chronic Disease Self-Management Program (CDSMP) is a group-based, 6-session, chronic disease self-management program largely focused on physical health self-management alone. I-IMR is delivered by community mental health providers or by community outreach workers, while CDSMP is co-delivered by two peers or by a health professional and a peer. Both programs have been widely recommended, disseminated, and used. The proposed parent study will randomize people with serious mental illness to I-IMR (n=300) and CDSMP (n=300).

The COVID-related Enhancement will involve enrolling 150 participants from the parent project to an evaluation of an additional I-IMR module compared to usual care during the pandemic. The I-IMR module will be delivered by trained interventionists in 3 calls over 3 weeks to n=75 I-IMR participants. The I-IMR participants and CDSMP participants will continue to receive Usual Care, consisting of generic support calls from clinicians at the study sites. Baseline, and 6, 9, and 12 week assessments will evaluate the effectiveness of the COVID-19 module that will be added to I-IMR.

ELIGIBILITY:
Inclusion Criteria:

* Serious Mental Illness (diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or chronic depression with moderate impairment in functioning) receiving services at Centerstone(KY and TN)
* Diagnosis of a chronic medical condition increasing risk of early mortality from cardiovascular or respiratory disease (e.g., diabetes, hyperlipidemia, hypertension, COPD, heart failure, tobacco dependence, obesity), and at least 1 ER visit or hospitalization within the past year or judgment by the treatment team of substantial need for illness self-management training.

Exclusion Criteria:

* Consumers who do not speak English
* Consumers with either no, or a well-controlled medical condition will not be included
* Individuals residing in a nursing home or other institution
* Evidence of significant cognitive impairment as indicated by a Mini Mental Status Examination score <24, will be excluded

Eligibility for the COVID -related substudy is dependent on enrollment and participation in the parent project (NCT03966872).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pratt, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Seven Counties Services, Louisville, Kentucky
  - Centerstone, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were actively participating in the parent project and maintained the randomization status from the parent study for the COVID intervention (see NCT03966870).
Period: Overall Study
Arm/Group | Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT: | Stanford Chronic Disease Self-Management Program (CDSMP) ONLY:
Started | 80 | 82
Completed | 77 | 80
Not Completed | 3 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT: | Stanford Chronic Disease Self-Management Program (CDSMP) ONLY: | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 80 | 158
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (9.9) | 49.1 (10.3) | 48.5 (10.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 26 | 21 | 47
  Female | 53 | 61 | 114
  Transgender/Other | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 28 | 57
  White | 40 | 48 | 88
  More than one race | 10 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received COVID-19 Vaccine
Description: change in status from baseline to follow up, receipt of vaccination or not.
Time Frame: Baseline to 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT: | Stanford Chronic Disease Self-Management Program (CDSMP) ONLY:
Number analyzed (Participants) | 80 | 82
Participants | 56 | 50

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Although All Cause Mortality was collected, serious adverse events were only collected when possibly/probably related to research participation
Arm/Group | Integrated Illness Management and Recovery (I-IMR) PLUS COVID-19 ENHANCEMENT: | Stanford Chronic Disease Self-Management Program (CDSMP) ONLY:
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/82
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/82
Other Adverse Events (participants affected / at risk) | 0/80 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05467982/Prot_SAP_000.pdf